CLINICAL TRIAL: NCT05520957
Title: Early Tracheostomy in COVID-19 Critically Ill Patients: A Retrospective Case Series
Brief Title: Early SARS-CoV-2 Tracheostomy
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital Zenica (Other)
Responsible Party: Principal Investigator, Mirza Kovacevic, Anesthesiologist, Cantonal Hospital Zenica
Other Study IDs: 4
Record Dates: First submitted 2022-08-28; First posted 2022-08-30 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Tracheostomy; Characteristics Disease; Metabolic Disturbance
Keywords: COVID-19; tracheostomy; demographic; lactate; D-dimer
MeSH Terms: conditions — COVID-19 | interventions — Tracheostomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tracheostomy — We collected data from all tracheotomised patients including age, sex, existing comorbidities, duration indicators (length of endotracheal intubation, day of tracheotomy, length of stay in the intensive care unit (ICU), and total length of hospital stay), respirator weaning marked with YES / NO. From the laboratory parameters, we analyzed: lactate, urea, creatinine, potassium and D-dimer. They were collected at two time intervals, before tracheotomy and after tracheotomy.

SUMMARY:
Objective of this case series was to evaluate the characteristics of early COVID-19 tracheostomy and its effect on laboratory parameters. A series of 17 patients with COVID-19undergo surgical tracheostomy in our intensive care unit. Demographic parameters, duration indicators, and laboratory parameters before and after tracheostomy were analyzed in patients. Of the 17 patients, 4 were men and 13 women with a mean age of 59 years. The average length of total hospitalization were 12 days, the length of stay in intensive care were 10 days, the length of endotracheal intubation were 9 days, with the seventh day of tracheotomy. Neurological and thyroid diseases and withdrawal had a statistically significant difference (p <0.05), with laboratory parameters without statistically difference. Critically ill COVID-19 patients undergoing early tracheostomy has a lower possibility of weaning from mechanical ventilation, and early tracheostomy itself has no significant effect on renal parameters, lactate and D-Dimer.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 postive patients
* surgery tracheostomy patients

Exclusion Criteria:

* trachestomy before admission in the ICU

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We performed a retrospective review of all COVID-19 critically ill patients who underwent tracheotomy between 2020 and 2022. All tracheotomized patients were included in the analysis, age 18 and older.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Characteristics of tracheotomized COVID-19 patients | 2 years
  We analysed age, sex, existing comorbidities, duration indicators (length of endotracheal intubation, day of tracheotomy, length of stay in the intensive care unit (ICU), and total length of hospital stay), respirator weaning marked with YES / NO. From the laboratory parameters, we analyzed: lactate, urea, creatinine, potassium and D-dimer. They were collected at two time intervals, before tracheotomy and after tracheotomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital, Zenica, Bosnia and Herzegovina